CLINICAL TRIAL: NCT02826148
Title: Validation of the French Adaptation of the Scale Aiding in the Diagnosis of the Autism Spectrum Disorders : Scale of Asperger Syndrome Diagnosis
Brief Title: Validation of the French Adaptation of the RAADS-R Scale : Scale of Asperger Syndrome Diagnosis
Acronym: RAADS-R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Fondation Orange (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8747
Record Dates: First submitted 2016-07-05; First posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-03

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with autism disorder (Other): The RAADS-R scale is a self-administered questionnaire completed by the patient himself assisted by a clinician
  Interventions: Other: RAADS-R scale

INTERVENTIONS:
Other: RAADS-R scale — This scale is a self-administered questionnaire completed by the person himself assisted by a clinician

SUMMARY:
The diagnosis of developmental disorders in adults is still difficult. Indeed, in France, there is not questionnaires to easily and accurately diagnose this disorder. Several diagnostic scales were developed in English. Among them, RAADS-R scale, which is a clinical tool that aims to better identify autism spectrum disorders including mild forms in adult people and help to diagnose of high-functioning autism . The objective of this study is to perform a complete validation of this scale in the french version.

DETAILED DESCRIPTION:
The diagnosis of developmental disorders in adults is still difficult. Indeed, in France, there is not questionnaires to easily and accurately diagnose this disorder. Several diagnostic scales were developed in English. Among them, RAADS-R scale, which is a clinical tool that aims to better identify autism spectrum disorders including mild forms in adult people and help to diagnose of high-functioning autism . This scale is a self-administered questionnaire completed by the person himself assisted by a clinician (psychiatrist, psychologist) which ensures the understanding of issues and the choice of answers. The scale contains 80 items including 64 questions describe specific symptoms of autism spectrum disorders and 16 questions describe non-symptomatic behaviors. The objective of this study is to perform a complete validation of this scale in the french version. 300 adults should be included, including 100 adults with high-functioning autism, 100 adults with another psychiatric disorder, and 100 adults without developmental disabilities and / or mental.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific criteria
* Collection of the informed consent (patient or legal representant)
* Affiliation or recipient with the mode of social security
* Current reading skills evaluated by completion of the fact sheet attached to the scale
* Age limits to > 18 years and < 75 years

Specific criteria

* Group of adult subjects with autism

  * Diagnosis of autism or Asperger syndrome established within the framework of a multidisciplinary evaluation (ADOS module 4 and/or ADI) using specific international classification criteria of rare diseases (CIM 10, DSM IV-R) (F84.0 et F84.5).
  * Intellectual efficiency estimated by means of a psychometric tool standardized (WAIS, WASI) greater than or equal to 85
  * Subjects not denying their symptoms
* Group of adult subjects with other psychiatric

  * Diagnosis of an other psychiatric trouble established according to the specific international classification criteria of mental diseases (CIM 10, DSM IV).
  * absence of pervasive developmental disorder diagnosis
  * Subjects not denying their symptoms
* Group of adult subjects not carriers of development and/or psychiatric disorders

Exclusion Criteria:

* Women pregnant and Breast-feeding
* Persons deprived of freedom by court order

Specific criteria

* Group of adult subjects with autism

  * Refusal of participation
  * absence of autism or Asperger syndrome diagnosis
* Group of adult subjects with other psychiatric

  * Refusal of participation
  * Pervasive developmental disorder diagnosis
* Group of adult subjects not carriers of development and/or psychiatric disorders

  * Refusal of participation
  * Diagnosis of cognitive development or psychomotor disorder, diagnosis of retard mental and/or psychiatric disorder.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2011-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
score at the RAADS-R scale | 15 days
  The scale contains 80 items including 64 questions describe specific symptoms of autism spectrum disorders and 16 questions describe non-symptomatic behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Amaria BAGHDADLI, MD-PhD, Principal Investigator — University Hospital, Montpellier

IPD SHARING:
Plan to Share IPD: No